CLINICAL TRIAL: NCT04909827
Title: 3D-printed Endocrowns Versus Prefabricated Zirconia Crowns for the Restoration of Pulpally-treated Primary Molars ; In-Vivo and In-Vitro Study
Brief Title: 3D-printed Endocrowns Versus Prefabricated Zirconia Crowns in Pulpally-treated Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lamia Hussein, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED 20-6D
Record Dates: First submitted 2021-05-26; First posted 2021-06-02 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Pulpotomy; Tooth Restoration
Keywords: 3D-printing; Endocrown; zirconia crown

STUDY DESIGN:
Intervention Model Description: A total of thirty primary mandibular molars in healthy subjects will be selected.
  The molars will be randomly assigned equally into two treatment groups
  1. Group A: 3D printed microfilled hybrid composite Endocrowns
  2. Group B: pr efabricated zirconia crowns Pulpotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): 3D printed microfilled hybrid composite Endocrowns
  Interventions: Procedure: 3D-printed endocrown
- group B (Experimental): prefabricated zirconia crowns
  Interventions: Procedure: Zirconia crown

INTERVENTIONS:
Procedure: 3D-printed endocrown — pulpotomy and restoration with 3D-printed microfilled hybrid composite endocrown
  Arms: group A
Procedure: Zirconia crown — pulpotomy and restoration with prefabricated zirconia crown
  Arms: group B

SUMMARY:
Aim of the study :

to compare between 3D printed microfilled hybrid composite endocrowns and prefabricated zirconia crowns for restoring pulpally treated primary molars regarding the following aspects: In Vivo aspects Patient satisfaction

*The esthetic, functional and biological performance according to FDI clinical criteria. At 3, 6 and 12 months

In Vitro aspects:

* Marginal gap.
* Fracture resistance.

Study methodology:

This study is a combined randomized clinical trial and in vitro study .The study will be conducted at the Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry,

Ain Shams University as follows:

In vivo comparison of the clinical performance of 3D printed Endocrowns versus prefabricated zirconia crowns regarding esthetic, functional and biological performance according to FDI clinical criteria. In vitro evaluation of the marginal gap and fracture resistance of both types of restorations.

DETAILED DESCRIPTION:
Study Procedure:

In-vivo Phase:

Study Population:

A total of thirty primary mandibular molars in healthy subjects will be selected from the Pediatric Dentistry and Dental Public Health outpatient clinic, Faculty of Dentistry, Ain Shams University. Randomization The molars will be assigned to one of the 2 groups using a generated computer list Allocation The molars will be allocated to the groups via a third party not involved with the study They will have the generated list and inform the allocation accordingly Blinding Is not possible due to the obvious difference between the 2 Pulpotomy procedure for both groups:

1. Local anesthesia will be administered.
2. Teeth will be isolated by a Rubber Dam.
3. Teeth will undergo pulpotomy procedure' as follows:

Caries will be removed using a large size 4 round bur, mounted onto a high speed hand piece with constant coolant. All access cavity walls are to be flared to allow complete exposure of the pulp chamber, and easy undisturbed access to the canals, followed by removal of all the soft pulpal tissue tags by a sharp spoon shaped excavator. Bleeding will be controlled using moist cotton pellet with gentle pressure. Formocresol will be applied through a cotton pellet for 5 mins, for fixation. The pulp chamber will be filled with reinforced zinc oxide and eugenol ( that will be mixed according to manufacturer s instructions. A 0.5 mm layer of Resin modified glass ionomer is then applied to the cavity floor and light cured for 40 secs, to isolate the zinc oxide eugenol paste, and block unwanted undercuts Analgesics will be prescribed to the patient to be taken when needed

Intervention :group A:

1. The cavities will be prepared so as to receive endocrowns:

   Occlusal preparation: achieved by drilling, 2mm depth grooves using diamond stone as guides for reduction of the occlusal surface. axial preparation: using a 7 degree taper diamond stone, eliminating undercuts in the access cavity.
2. impression for the preparation is taken using putty and light poly vinyl siloxane material
3. Light cured temporary filling will be placed in the cavity as temporisation.
4. The impression will be sent to the lab and the patient is dismissed
5. The preparation will be optically scanned in the lab and the restoration will be digitally designed using computer designing software.
6. The restoration will be printed using 3D printer using microfilled hybrid composite material.
7. During the second visit the temporary is removed the restoration is cemented by self adhesive resin after etching and bonding the cavity.

Control Group B:

1. Crown reduction:

   reduction will be performed on the occlusal surface disregarding the occlusal anatomy using a flame stone or a wheel stone, to perform occlusal clearance. Then reduction will be performed on the mesial, distal, buccal and lingual surfaces of the tooth to compensate for the thickness of the zirconia crowns. Reduction will first be performed using fine needle stone to free the contact from the adjacent teeth then followed by reduction of the other surfaces using a diamond stone. Roundation of the line angles will be performed
2. Zirconia crowns that match the size of the tooth will be selected putting into consideration that no undercuts should be present to avoid crown fracture.
3. . After checking the size of the crowns, it will be removed, drie d and cemented on the tooth using (3M™ ESPE™ KETAC™ CEM) that will be mixed according to manufacturer's instructions.
4. Pressure will be applied on the crown, and any excess cement will be removed after it hardens. All children and parents will be give n strict oral hygiene instructions and dietary instructions Teeth not included in the study will be scheduled for dental treatment in the Department of Pediatric Dentistry, Faculty of Dentistry, Ain Shams University. Outcome measurement

Esthetic functional biological criteria will be evaluated in the following order:

After cementation evaluation: patients will be evaluated according to FDI criteria as previously mentioned,.

In Vitro phase:

All soft tissue debris will be removed by a hand scaler and teeth will be disinfect ed, and then stored in distilled water at 4 degrees Celsius until the start of the study.

The molars will undergo pulpotomy procedures and filled as previously described. The molars will be randomly divided into two groups Group A: Will receive 3D printed Endocrowns Group B: Will receive prefabricated zirconia crowns The specimens will be embedded perpendicularly in Polyvinyl chloride ( cubes with the occlusal surface parallel to the ground using acrylic resin extending 2mm b elow the cemento enamel junction. The following will be measured: Marginal gap Precementation measurements of the cervical vertical marginal discrepancies will be performed before cementation. For each specimen, four stereomicrographs will be captured by a stereomicroscope (Wild 400, Switzerland) at a 32× magnification. Images will then be transferred to the computer software for image analysis

Fracture Resistance:

An axial loading condition through the functional cusp will be defined in the mechanical failure description. Failure to fracture strength will be tested with a universal testing machine at a 0.5 mm/sec crosshead speed. Application of a round end vertical loading tip on the occlusal third of a specimen fixed into a loading apparatus as functional loading simulation.

Data Management:

Patient information will be gathered and stored in the patient examination chart of the outpatient clinic, Department of Pediatric Dentistry, faculty of Dentistry, Ain Shams University. All information will be kept as a hard copy and as an electronic one as well. Patient information will be guarded as co nfidential information that should never be revealed at all times. This file will remain with the investigator during the study.

Statistical Analysis:

All data will be tabulated, summarized and statistically analyzed using software SPSS (Statistical Packages for Social Sciences. 3 and 6 months evaluation: evaluation of the previous criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Having at least one vital primary molar with deep carious lesion indicated for pulpotomy or pulpectomy.
2. The anticipated exfoliation date of the selected primary teeth has to be more than 12 months from the date of the study start.

Exclusion criteria:

1. Children who are uncooperative needing sedatin or general anasthesia.
2. Children who are physically or mentally disabled or having any medical condition that will complicate the treatment.

e) Teeth of poor prognosis due to th e presence of an abscess or a sinus, mobility, advanced bone or root resorption.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
clinical performance | 6 months
  Federation Dentaire international clinical assessment scale. Minimum value is 1 and highest value is 11. Higher values mean worst outcome.

SECONDARY OUTCOMES:
patient satisfaction | 6 months
  A structured patient satisfaction questionnaire with a 3 points likert scale question.

CONTACTS AND LOCATIONS:
Overall Officials: Mariem O Wassel, PhD, Study Director — Ainshams university
Locations (1):
- Ain shams university, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbas LH, Wassel MO, Hassan IT, El-Dimeery AG, Elghazawy RK. 3D printed endocrowns versus prefabricated zirconia crowns for pulpotomized primary molars: A randomized controlled trial. J Dent. 2025 Feb;153:105556. doi: 10.1016/j.jdent.2025.105556. Epub 2025 Jan 6. PMID 39778737